CLINICAL TRIAL: NCT02078518
Title: Level of Physical Activity and Its Associations With Fatigue and Quality of Life in Multiple Myeloma Survivors
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Principal Investigator, Haematology-Oncology, Chng Wee Joo, National University Hospital, Singapore
Other Study IDs: 2013/00724
Record Dates: First submitted 2013-12-09; First posted 2014-03-05 (Estimated); Last update posted 2014-03-05 (Estimated); Status verified 2014-03

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Multiple Myeloma: Questionnaires will be given to patients for completion.
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires

SUMMARY:
The purpose of this study is to gives understanding to level of physical activity, occurrence of fatigue and quality of life amongst multiple myeloma survivors in the local setting. As multiple myeloma survival improves, it is vital to focus on interventions that will help to maximize QOL. A positive correlation may suggest that exercise is such an intervention.

The hypothesis are multiple myeloma survivors are performing low levels of physical activity. Higher levels of physical activity will be associated with higher levels of QOL and lower fatigue levels.

DETAILED DESCRIPTION:
Multiple myeloma its associated treatment often result in persistent symptoms such as fatigue, pain, neuropathy and diminished functional performance that can affect the survivor's quality of life (QOL). And as survival for multiple myeloma continues to improve, physical activity may be a supportive therapy that can help to address the multitude of QOL concerns. Physical activity is a modifiable behavior, and has been proposed as an important non-pharmacologic intervention to improve health-related outcomes among cancer survivors. The American College of Sports Medicine examined evidence of the impact of physical activity in cancer survivors, and concluded that physical activity is safe for cancer patients, both during and after cancer treatment, and may lead to improved physical functioning, decreased physical fatigue, and improved QOL in a number of cancer survivor groups, including hematopoietic malignancies. While a small number of studies have suggested that exercise may reap benefits in QOL and fatigue in multiple myeloma survivors, none were conducted in the local context.Given the limited evidence, the primary objectives of this preliminary study is to estimate the prevalence of physical activity among a local sample of multiple myeloma survivors, and to investigate its associations with reported fatigue and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Multiple Myeloma
* Able to complete questionnaires

Exclusion Criteria:

- Unable to complete questionnaires

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Multiple Myeloma patients treated in National University Hospital.
Sampling Method: Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2013-09; Primary Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
Change in the level of physical activity, occurrence of fatigue and quality of life amongst multiple myeloma survivors in the local setting | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- National University Hospital, Singapore, Singapore

REFERENCES:
- [Background] Jones LW, Courneya KS, Vallance JK, Ladha AB, Mant MJ, Belch AR, Stewart DA, Reiman T. Association between exercise and quality of life in multiple myeloma cancer survivors. Support Care Cancer. 2004 Nov;12(11):780-8. doi: 10.1007/s00520-004-0668-4. PMID 15322968
- [Background] Coleman EA, Goodwin JA, Coon SK, Richards K, Enderlin C, Kennedy R, Stewart CB, McNatt P, Lockhart K, Anaissie EJ, Barlogie B. Fatigue, sleep, pain, mood, and performance status in patients with multiple myeloma. Cancer Nurs. 2011 May-Jun;34(3):219-27. doi: 10.1097/NCC.0b013e3181f9904d. PMID 21522061